CLINICAL TRIAL: NCT01718197
Title: Clinical and Molecular Phenotypes of Severe Asthma
Brief Title: Severe Asthma Research Program (SARP)- San Francisco Clinical Site
Acronym: SARP
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: SARP-SF; 5U10HL109146-04 (NIH)
Record Dates: First submitted 2012-10-27; First posted 2012-10-31 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Severe Asthma; Bronchoscopy
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood: CBC/Diff, Total IgE, Serum, Plasma, DNA, RNA Urine EBC Sputum: Supernatant, Cell Pellet Bronchoscopy: BAL, Bronchial Brushings, Bronchial Biopsy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Mild-to-Moderate Asthma: Those with mild-to-moderate persistent asthma as defined by the NAEPP EPR-3 guidelines.
- Severe Asthma: Major Criteria: (1 required)
  1. Treatment with oral corticosteroids for at least 6 of the previous 12 months
  2. Treatment with high-dose inhaled corticosteroids (ICS) for at least 10 of the previous 12 months
  Minor Criteria: (2 required)
  1. Daily treatment with an asthma controller medication in addition to ICS, or
  2. Asthma symptoms requiring short-acting bronchodilator use on a daily or near daily basis, or
  3. Persistent airway obstruction with baseline FEV1 <80% predicted, or
  4. ≥ 1 urgent visits for asthma in the previous 12 months, or
  5. ≥ 3 systemic corticosteroid bursts in the previous 12 months, or
  6. Prompt deterioration with a reduction in oral or inhaled corticosteroid dose, or
  7. A near-fatal asthma event (i.e., intubation) in the past
- Healthy Controls: Those without asthma or other chronic lung disease.

SUMMARY:
The mission of SARP is to improve the understanding of severe asthma through integrated study of its clinical and biological features and to evaluate their changes over time. The ultimate goal of these efforts is to promote better treatments for severe asthma.

DETAILED DESCRIPTION:
The mission of the SARP is to improve the understanding of severe asthma to develop better treatments. The SARP will gain a better understanding of asthma and its endotypes, in children and adults, by defining the disease at the molecular and cellular levels in the context of the temporal phenotypic expression of the disease. To this end, the SARP investigators will utilize both mechanistic and evoked phenotype approaches to: 1) characterize developmental molecular, cellular and physiologic phenotypes in children and adults with mild to severe asthma, and 2) to further elucidate the evolving pathobiology and pathogenesis of severe asthma and its sub-phenotypes and 3) compare these features over time.

This approach involves a shared longitudinal protocol conducted across all participating centers which includes common information on all SARP participants. Additionally, the SARP-SF has identified mechanistic research questions to be included in the shared longitudinal protocol. This will be explored through additional sample collections of sputum and fluids and biopsied tissue collected by bronchoscopy. Together, these longitudinal and mechanistic approaches will enable prediction of phenotype stability/fluctuation and pharmacologic responses and identification of novel, disease-modifying targets for treatment.

ELIGIBILITY:
Inclusion Criteria:

* FEV1 bronchodilator reversibility ≥12% or airway hyperresponsiveness reflected by a methacholine PC20 ≤16 mg/mL
* An exception will be made for enrollees whose FEV1 is < 50% predicted (<70% in children aged 6 to 17 years), precluding methacholine challenge testing. If bronchodilator reversibility is <12% in these participants, a diagnosis of asthma acceptable to the investigator is sufficient for inclusion in SARP.

Exclusion Criteria:

* Pregnancy during the characterization phase,
* Current smoking,
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age,
* Other chronic pulmonary disorders associated with asthma-like symptoms, including (but not limited to) cystic fibrosis, chronic obstructive pulmonary disease, chronic bronchitis, vocal cord dysfunction (that is the sole cause of respiratory symptoms and at the PI's discretion), severe scoliosis or chest wall deformities that affect lung function, or congenital disorders of the lungs or airways,
* History of premature birth before 35 weeks gestation,
* Unwillingness to receive an intramuscular triamcinolone acetonide injection
* Evidence that the participant or family may be unreliable or poorly adherent to their asthma treatment or study procedures,
* Planning to relocate from the clinical center area before study completion,
* Any other criteria that place the subject at unnecessary risk according to the judgment of the Principal Investigator and/or attending physician(s) of record, or
* Currently participating in an investigational drug trial.

Healthy Controls:

Inclusion criteria: Healthy subjects between the age of 18y and 65y. At least 3 of the 7 subjects per center should be aged 35y or older.

Exclusion criteria

* History of chronic diseases that affect the lungs.
* A history suggestive of allergic rhinitis, eczema or chronic sinusitis.
* An improvement in FEV1 of more than 12% following 4 puffs of albuterol.
* Smoking history > 10 pack years if ≥30 years of age, or smoking history > 5 pack years if <30 years of age, or any smoking within the past year.
* Respiratory tract infection within the past 4 weeks.
* Pregnancy.
* History of premature birth (<35 weeks).

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A diverse sample of subjects with asthma is needed to gain better understanding of asthma and its endotypes. SARP will therefore enroll subjects 6 years and older with a physician diagnosis of asthma. The target recruitment goal for each center is 75% adults (age 18 and older) and 25% children age 6-17 years. Within the pediatric age group, an attempt will be made to enroll equal numbers of children 6-11 and 12-17 years of age. Similarly, an attempt will be made to enroll at least 50% females and 30% minorities.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2020-02-18 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Lung function decline | Enrollment, 1 year, 2 years, 3 years
  Changes in lung function parameters over time.

SECONDARY OUTCOMES:
Exacerbation frequency | Monthly for 3 years
  Number of oral corticosteroid requiring exacerbations of asthma
Inflammatory cellular markers | Enrollment, 1 year, 2 years, 3 years
  Changes in inflammatory cellular markers in sputum, exhaled breath, and blood.

CONTACTS AND LOCATIONS:
Overall Officials: John V Fahy, MD, MSc, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Huang BK, Elicker BM, Henry TS, Kallianos KG, Hahn LD, Tang M, Heng F, McCulloch CE, Bhakta NR, Majumdar S, Choi J, Denlinger LC, Fain SB, Hastie AT, Hoffman EA, Israel E, Jarjour NN, Levy BD, Mauger DT, Sumino K, Wenzel SE, Castro M, Woodruff PG, Fahy JV, Sarp FTNSARP. Persistent mucus plugs in proximal airways are consequential for airflow limitation in asthma. JCI Insight. 2024 Feb 8;9(3):e174124. doi: 10.1172/jci.insight.174124. PMID 38127464
- [Derived] Dunican EM, Elicker BM, Gierada DS, Nagle SK, Schiebler ML, Newell JD, Raymond WW, Lachowicz-Scroggins ME, Di Maio S, Hoffman EA, Castro M, Fain SB, Jarjour NN, Israel E, Levy BD, Erzurum SC, Wenzel SE, Meyers DA, Bleecker ER, Phillips BR, Mauger DT, Gordon ED, Woodruff PG, Peters MC, Fahy JV; National Heart Lung and Blood Institute (NHLBI) Severe Asthma Research Program (SARP). Mucus plugs in patients with asthma linked to eosinophilia and airflow obstruction. J Clin Invest. 2018 Mar 1;128(3):997-1009. doi: 10.1172/JCI95693. Epub 2018 Feb 5. PMID 29400693
- See also: Severe Asthma Research Program Main Webpage — http://www.severeasthma.org/
- See also: UCSF Recruitment Website — http://acrc.ucsf.edu/